CLINICAL TRIAL: NCT05837442
Title: The Effect Of Osteopathic Manual Therapy On Arterial Circulation In Patients With Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Muhammet Ayhan ORAL, Assistant Professor, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OMT on PAD
Record Dates: First submitted 2023-04-06; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Peripheral Arterial Disease; Osteopathy in Diseases Classified Elsewhere
Keywords: peripheral arterial disease; osteopathic manual therapy; artery diameter; arterial flow
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: 28 Patients were included. All of the patients included in the study were informed about the process. Voluntary consent was obtained from the patients participating in the study. 14 of the patients were randomly assigned to the osteopathic manual therapy group (OMTG) and 14 to the control group (CG).
Who Masked: Participant, Investigator
Masking Description: In this double-blind study, the physician who performed the radiological evaluation was unaware of which group the individual belonged to, and the patients were unaware of which group they belonged to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic Manual Therapy Group (OMTG) (Experimental): The total duration of all techniques applied is 30 minutes. The techniques used in the extremities were applied to both extremities.
  Interventions: Other: Osteopathic Manual Therapy
- Control Group (CG) (No Intervention): No intervention was made to the patients in the control group.

INTERVENTIONS:
Other: Osteopathic Manual Therapy — Occipital release, supraclavicular release, sternum mobilization, omentum minus release, liver pumping, diaphragm mobilization, grand maneuver for 3 minutes, general osteopathic manual therapy of the hip, knee and ankle was applied to each extremity for 90 seconds for a total of 3 minutes
  Arms: Osteopathic Manual Therapy Group (OMTG)

SUMMARY:
Peripheral artery disease (PAD) is a chronic atherosclerotic process that causes narrowing of peripheral arterial vessels in the lower extremities. Osteopathic manual therapy (OMT) is one of the new treatment options for various pathologies. The aim of this study was to investigate the effect of OMT on arterial circulation in patients with PAD.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is a chronic, atherosclerotic process in the lower extremities that causes narrowing of the peripheral arteries. It has a prevalence of up to 10% worldwide, this rate rises to about 30% in patients over 50 years of age. Atherosclerosis is characterized by intimal lesions called atheromas or atheromatous or fibrous fatty plaques that protrude into the vascular lumen, weakening the underlying environment. In atherosclerotic disease of the lower extremities, arterial stenoses cause a gradual reduction of prolonged blood flow, which manifests clinically as pain and tissue loss. Many patients with PAD are asymptomatic. The earliest symptom of the disease is pain while walking and is known as intermittent claudication (IC). If IC left untreated, it can cause pain at rest, tissue loss, or gangrene. Risk factors for peripheral arterial disease can be listed as age, gender, ethnicity, smoking, diabetes, hypertension, hyperlipidemia, chronic kidney failure. Understanding the underlying pathophysiological mechanisms of atherosclerosis and the finding of intermittent claudication in PAD is essential to be aware of the whole process and recommend prevention and treatment strategies. Patients with a diagnosis of PAH should receive a comprehensive treatment program, including structural exercise and lifestyle modification, to reduce cardiovascular ischemic events and improve functional status. All treatment plans should include aggressive modification of risk factors. This includes smoking cessation, weight loss, diet, hyperlipidemia, hypertension, diabetes, homocysteine, inflammation, antiplatelet medication, exercise. Recently, manual therapy methods have also been used.

Andrew Taylor Still, founder of osteopathic manual therapy (OMT), was born on August 6, 1828, in Jonesville. He developed a strong belief in God as the perfect creator of all things. Because of this, he had the belief that all creation, including the human body, is perfect. He stated that a perfect body can heal itself and will contain the necessary tools for this. In OMT, 5 models are used to treat the person: biomechanic, respiratory-circulatory, metabolic-energy, neurological and behavioral. The circulatory model is concerned with the maintenance and enhancement of the extracellular environments through the delivery of oxygen and nutrients and the removal of cellular waste products. In this model, the clinical goal is to identify and eliminate key tissue stresses that impede the flow or circulation of body fluids to positively impact tissue health. The circulatory model is one of three levers used in the treatment of systemic dysfunction. In this model, coordinated OMT allows to improve homeostasis. These effects are known to be caused by nitric oxide (NO). Salomon et al. concluded that mechanical stimulation of excised neural and vascular tissue stimulates NO release, based on the data they obtained in their laboratory. Stimulation of muscle structure within physiological limits by manual techniques causes NO synthase enzyme activation, followed by NO release in a short time. The effect of NO, which is released in a short time, can cause a longer-term physiological mechanisms, especially in vascular structures. NO regulates by reducing endothelial and immunocyte activation and adhesion, thereby performing vital physiological activities including vasodilation. This can act as a positive feedback mechanism that causes the amount of blood flow to increase. As a result of NO-induced vasodilation, the organism has the potential to protect itself from microorganisms and physiological disorders such as hypertension. Vasodilation modulated by NO also reduces endothelial dysfunction. There are studies in the literature reporting that manual therapy interventions contribute to the systemic circulation, but only one study in which OMT was applied in patients with PAH was found. In this study, patients' ABI, functional performance, quality of life and some blood parameters were evaluated. No data was performed on arterial diameter and flow in the affected extremity. Considering the NO-induced vasodilator effects of OMT, it can be thought that it may increase circulation and change arterial diameter and flow in patients with PAD. Purpose of this study, to investigate the effect of osteopathic manual therapy on arterial circulation in patients with PAD.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with PAD,
* clinical onset of the disease for at least 3 months,
* ABI value between 0.4 and 1.4,
* Grade 2b according to Fontaine classification system,

Exclusion Criteria:

* vascular or endovascular surgery in the last 3 months,
* unstable angina,
* myocardial infarction (MI),
* stroke,
* heart failure,
* significant hepatic or renal failure (dialysis-related etc.),
* acute infectious disease,
* neoplasia

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Femoral Artery Diameter Doppler Ultrasonography | 10 minutes
  Femoral artery diameter evaluated by radiologist. The femoral artery diameter unit is in mm (millimeters).
  In the evaluation, the wall contour characteristics of the vessel to be examined were evaluated and the diameter was measured.
Femoral Artery Flow Doppler Ultrasonography | 10 minutes
  Femoral artery flow evaluated by radiologist. The femoral artery flow unit is in ml/sn (milliliter/second).
  Peak systolic and end diastolic flow rates were measured by spectral examination
Six minute walk test | 6 minutes
  The six minute walk test unit is in m(meter)
  During the test, the patient is asked to walk as fast as he can without running, and the total distance he/she walks is measured after 6 minutes. The walking area must be at least 30 m long. Standardized warnings are used during testing. The test is terminated immediately in case of chest pain, intolerable dyspnea, leg cramps, extreme tiredness, sweating and pallor. It is possible to stop and rest during the test. As a result of the test, the total distance walked by the patient after six minutes was recorded

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMET AYHAN ORAL, Principal Investigator — Kırıkkale University
Locations (1):
- Kirikkale University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group; Bell K, Caporusso J, Durand-Zaleski I, Komori K, Lammer J, Liapis C, Novo S, Razavi M, Robbs J, Schaper N, Shigematsu H, Sapoval M, White C, White J, Clement D, Creager M, Jaff M, Mohler E 3rd, Rutherford RB, Sheehan P, Sillesen H, Rosenfield K. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). Eur J Vasc Endovasc Surg. 2007;33 Suppl 1:S1-75. doi: 10.1016/j.ejvs.2006.09.024. Epub 2006 Nov 29. No abstract available. PMID 17140820
- [Background] Mascarenhas JV, Albayati MA, Shearman CP, Jude EB. Peripheral arterial disease. Endocrinol Metab Clin North Am. 2014 Mar;43(1):149-66. doi: 10.1016/j.ecl.2013.09.003. PMID 24582096
- [Background] Kannel WB, Wilson PW. An update on coronary risk factors. Med Clin North Am. 1995 Sep;79(5):951-71. doi: 10.1016/s0025-7125(16)30016-5. PMID 7674694
- [Background] Hiatt WR, Armstrong EJ, Larson CJ, Brass EP. Pathogenesis of the limb manifestations and exercise limitations in peripheral artery disease. Circ Res. 2015 Apr 24;116(9):1527-39. doi: 10.1161/CIRCRESAHA.116.303566. PMID 25908726
- [Background] Conte SM, Vale PR. Peripheral Arterial Disease. Heart Lung Circ. 2018 Apr;27(4):427-432. doi: 10.1016/j.hlc.2017.10.014. Epub 2017 Nov 7. PMID 29150158
- [Background] Degenhardt BF, Kuchera ML. Update on osteopathic medical concepts and the lymphatic system. J Am Osteopath Assoc. 1996 Feb;96(2):97-100. doi: 10.7556/jaoa.1996.96.2.97. PMID 8838905
- [Background] Backer M, Hammes MG, Valet M, Deppe M, Conrad B, Tolle TR, Dobos G. Different modes of manual acupuncture stimulation differentially modulate cerebral blood flow velocity, arterial blood pressure and heart rate in human subjects. Neurosci Lett. 2002 Nov 29;333(3):203-6. doi: 10.1016/s0304-3940(02)01109-6. PMID 12429383
- [Background] Salamon E, Zhu W, Stefano GB. Nitric oxide as a possible mechanism for understanding the therapeutic effects of osteopathic manipulative medicine (Review). Int J Mol Med. 2004 Sep;14(3):443-9. PMID 15289898
- [Background] Stefano GB, Goumon Y, Bilfinger TV, Welters ID, Cadet P. Basal nitric oxide limits immune, nervous and cardiovascular excitation: human endothelia express a mu opiate receptor. Prog Neurobiol. 2000 Apr;60(6):513-30. doi: 10.1016/s0301-0082(99)00038-6. PMID 10739087
- [Background] Walkowski S, Singh M, Puertas J, Pate M, Goodrum K, Benencia F. Osteopathic manipulative therapy induces early plasma cytokine release and mobilization of a population of blood dendritic cells. PLoS One. 2014 Mar 10;9(3):e90132. doi: 10.1371/journal.pone.0090132. eCollection 2014. PMID 24614605
- [Background] Lombardini R, Marchesi S, Collebrusco L, Vaudo G, Pasqualini L, Ciuffetti G, Brozzetti M, Lupattelli G, Mannarino E. The use of osteopathic manipulative treatment as adjuvant therapy in patients with peripheral arterial disease. Man Ther. 2009 Aug;14(4):439-43. doi: 10.1016/j.math.2008.08.002. Epub 2008 Sep 27. PMID 18824395
- [Background] Noll DR. Short-term hematologic and hemodynamic effects of osteopathic lymphatic techniques. J Am Osteopath Assoc. 2009 Mar;109(3):121-2; author reply 122-3. No abstract available. PMID 19336762
- [Background] Kilgore T, Malia M, Di Giacinto B, Minter S, Samies J. Adjuvant Lymphatic Osteopathic Manipulative Treatment in Patients With Lower-Extremity Ulcers: Effects on Wound Healing and Edema. J Am Osteopath Assoc. 2018 Dec 1;118(12):798-805. doi: 10.7556/jaoa.2018.172. PMID 30476991